CLINICAL TRIAL: NCT03667807
Title: Transcranial Magnetic Stimulation (TMS)-Induced Plasticity Improving Cognitive Control in Obsessive-compulsive Disorder (OCD)
Brief Title: TMS-induced Plasticity Improving Cognitive Control in OCD
Acronym: TIPICCO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, O.A. van den Heuvel, Professor of Neuropsychiatry, Amsterdam UMC, location VUmc
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 91717306
Record Dates: First submitted 2018-09-06; First posted 2018-09-12 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Obsessive-Compulsive Disorder
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- rTMS condition 1 (Experimental)
  Interventions: Device: Repetitive transcranial magnetic stimulation
- rTMS condition 2 (Experimental)
  Interventions: Device: Repetitive transcranial magnetic stimulation
- rTMS condition 3 (Experimental)
  Interventions: Device: Repetitive transcranial magnetic stimulation

INTERVENTIONS:
Device: Repetitive transcranial magnetic stimulation — Non invasive brain stimulation
  Other Names: rTMS, TMS

SUMMARY:
Repetitive transcranial magnetic stimulation (rTMS) has been shown in several previous clinical trials to be an effective treatment for obsessive-compulsive disorder (OCD). However, the neural working mechanisms of rTMS in OCD are unknown, and the optimal stimulation sites have not yet been established. Our study aims to compare the clinical and neurobiological effects of three different rTMS stimulation protocols in OCD patients. 8 weeks of rTMS therapy will be delivered in combination with cognitive behavioural therapy. Multimodal neuroimaging will be carried out before and after treatment in order to demonstrate the neurobiological effects of the therapy.

ELIGIBILITY:
Inclusion Criteria:

OCD patients:

* Age between 18 and 65
* Primary DSM-5 diagnosis of OCD
* Moderate to severe OCD symptoms (expressed as a minimum score of 16 on the Yale - Brown Obsessive Compulsive Scale (YBOCS)
* Unmedicated or stable dose of medication for at least 12 weeks prior to randomisation - with no plans to change dose during the study period
* At least 1 previous attempt at cognitive behavioural therapy (CBT) in lifetime
* At least 1 previous attempt with serotonergic medication or strong preference for non-pharmacological treatment
* Capacity to provide informed consent

Healthy controls (baseline measurements only):

* Age between 18 and 65
* Capacity to provide informed consent

Exclusion Criteria:

OCD patients:

* MRI exclusion criteria (metal in body, pregnancy)
* TMS exclusion criteria (metal in body, history of epilepsy)
* Schizophrenia, bipolar disorder, active suicidal ideation, use of antipsychotics within last 12 weeks
* previous experience with rTMS as treatment

Healthy controls:

* Current Diagnostic and Statistical Manual (DSM)-5 diagnosis
* Personal history of DSM-5 diagnosis
* use of psychotropic medications within last 12 months
* 1st degree family member with OCD
* MRI exclusion criteria (as above)
* TMS exclusion criteria (as above)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2019-05-08 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
task based functional magnetic resonance imaging (fMRI) blood oxygen level dependent (BOLD) response | Baseline and 12 weeks (i.e. post-treatment)
  Change in task based fMRI BOLD response following rTMS

SECONDARY OUTCOMES:
Yale-Brown Obsessive Compulsive Scale (Y-BOCS) | Baseline, 6 weeks, (i.e. during treatment), 12 weeks (i.e. post-treatment), 22 weeks (i.e. follow-up)
  OCD symptom severity

OTHER OUTCOMES:
Functional connectivity | Baseline and 12 weeks (i.e. post-treatment)
  Measured using resting state fMRI
Structural connectivity | Baseline and 12 weeks (i.e. post-treatment)
  Measured using diffusion tensor imaging (DTI) MRI
Cortical excitation and inhibition (Motor-evoked potential amplitude, TMS-evoked potential, short interval cortical inhibition, long interval cortical inhibition) | Baseline, 6 weeks, (i.e. during treatment), 12 weeks (i.e. post-treatment), 22 weeks (i.e. follow-up)
  Measured using single and double pulse TMS + electromyography (EMG) / electroencephalography (EEG)
Neurotransmitter concentrations | Baseline and 12 weeks (i.e. post-treatment)
  Measured using magnetic resonance spectroscopy (MRS)
Planning | Baseline, 12 weeks (i.e. post-treatment)
  Measured using Tower of London cognitive task
Response inhibition | Baseline, 12 weeks (i.e. post-treatment)
  Measured using the stop-signal cognitive task
Error processing | Baseline, 6 weeks, (i.e. during treatment), 12 weeks (i.e. post-treatment), 22 weeks (i.e. follow-up)
  Measured using the Flanker cognitive task
EEG measures | Baseline, 6 weeks, (i.e. during treatment), 12 weeks (i.e. post-treatment), 22 weeks (i.e. follow-up)
  Resting state EEG, EEG event related potentials measured during tasks (Error related negativity using Flanker task, Late Positive Potential during appraisal of emotional stimuli)

CONTACTS AND LOCATIONS:
Locations (1):
- Amsterdam UMC, location VU Medical Center, Amsterdam, North Holland, Netherlands

REFERENCES:
- [Derived] Fitzsimmons SMDD, Postma T, van Campen AD, Vriend C, Batelaan NM, van Oppen P, Hoogendoorn AW, van der Werf YD, van den Heuvel OA. TMS-induced plasticity improving cognitive control in OCD I: Clinical and neuroimaging outcomes from a randomised trial of rTMS for OCD. medRxiv [Preprint]. 2023 Nov 5:2023.11.04.23298100. doi: 10.1101/2023.11.04.23298100. PMID 37961433